CLINICAL TRIAL: NCT04003012
Title: Pain Control in Pediatric Oncology: Utility of EMLA Cream vs Lidocaine Injection in Lumbar Punctures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Mohamad Badawi, MD, Assistant Professor WVU-Charleston, CAMC Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-567
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Leukemia-Lymphoma
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EMLA (Active Comparator): The patient will receive 5 grams EMLA cream at the site of the lumbar puncture at least 60 minutes prior to procedure. The site of EMLA application will be covered with Tegaderm dressing.
  Interventions: Drug: EMLA
- Lidocaine (Active Comparator): The patient will receive sham-EMLA cream (a fragrance-free hypoallergenic moisturizer cream) will be applied at least 60 minutes per standard protocol with Tegaderm dressing.- Following conscious sedation, the patient will receive lidocaine 1% injection (~1-2ml) at the appropriate site 30-60 seconds prior to LP needle insertion.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: EMLA — EMLA cream (lidocaine 2.5% and prilocaine 2.5%)
  Arms: EMLA
Drug: Lidocaine — lidocaine 1%
  Arms: Lidocaine

SUMMARY:
A common procedure in children with cancer is the spinal tap, or lumbar puncture (LP), in which a needle is inserted into the spinal canal. In this population, LPs are most commonly performed to collect cerebrospinal fluid (CSF, the liquid surrounding the brain and spinal cord) for diagnostic testing, and to inject medications including chemotherapy. Local analgesic (pain control medicine) during pediatric LP procedures is underutilized and not standardized. The first local analgesic routinely used for LP procedures was lidocaine injection. The discovery of the topical EMLA (lidocaine 2.5%/prilocaine 2.5%) cream, approved by the FDA for local skin use in pediatric patients, has provided an additional option for local LP analgesia. A comparison between topical EMLA vs lidocaine injection for LP pain control in the pediatric population has not been performed. Pediatric oncology patients often require serial LPs for diagnostics purposes and/or chemotherapy delivery. Due to a lack of standardization of LP analgesia in this population, the investigators have designed a prospective, single-blind, randomized control crossover trial to examine EMLA vs. lidocaine injection in reducing pain associated with LP in children being treated for leukemia or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cancer patients (aged 3-18) with a diagnosis of leukemia or lymphoma
* Patients are expected to receive serial (i.e. > 1) LP as outpatients in Charleston Area Medical Center Children's Cancer Center in the course of 12 months for diagnostic and/or treatment purposes

Exclusion Criteria:

* Patients not in the age range
* Non-cancer patients
* Allergy to amide anesthetics
* Patients treated with class I and III anti-arrhythmic drugs (eg, amiodarone, bretylium, sotalol, dofetilide)
* Patients with congenital or idiopathic methemoglobinemia

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Badawi, MD, Principal Investigator — WVU-Charleston and CAMC
Locations (1):
- CAMC - Women and Children's Hospital, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients were screen and enrolled in the study
Groups:
- EMLA for First Lumbar Puncture, Lidocaine Injection for Second Lumbar Puncture: First lumbar puncture: the participant received 5 grams EMLA cream at the site of the lumbar puncture at least 60 minutes prior to procedure.
  Subsequent lumbar puncture: patient received sham-EMLA cream applied at least 60 minutes prior to procedure. Following conscious sedation, the patient received lidocaine 1% injection (~1-2ml) 30-60 seconds prior to lumbar puncture needle insertion.
- Lidocaine Injection for First Lumbar Puncture, EMLA for Second Lumbar Puncture: First lumbar puncture: patient received sham-EMLA cream applied at least 60 minutes prior to procedure. Following conscious sedation, the patient received lidocaine 1% injection (~1-2ml) 30-60 seconds prior to lumbar puncture needle insertion. the participant received 5 grams EMLA cream at the site of the lumbar puncture at least 60 minutes prior to procedure.
  Subsequent lumbar puncture: the participant received 5 grams EMLA cream at the site of the lumbar puncture at least 60 minutes prior to procedure.
Period: Overall Study
Arm/Group | EMLA for First Lumbar Puncture, Lidocaine Injection for Second Lumbar Puncture | Lidocaine Injection for First Lumbar Puncture, EMLA for Second Lumbar Puncture
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMLA for First Lumbar Puncture, Lidocaine Injection for Second Lumbar Puncture | Lidocaine Injection for First Lumbar Puncture, EMLA for Second Lumbar Puncture | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [3.5 to 14] | 6 [4 to 11] | 5.5 [4 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Post Lumbar Puncture Pain: Wong-Baker Faces Pain Rating Scale
Description: Pain was self-reported by the child using the validated pain scale, Wong-Baker Faces Pain Rating Scale. The scale shows a series of six faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain, with higher the number, greater the pain.
  Below are the median and range of values (minimal to maximal) reported by each arm's 10 patients. Reported values were identical between arms.
Time Frame: , pain will be assessed at 30 - 60 minutes after waking up after lumbar puncture and 24 hours after lumbar puncture
Measure: Median (Full Range); unit: score on a scale
Groups:
- EMLA: Participants who received 5 grams EMLA cream at the site of the lumbar puncture at least 60 minutes prior to procedure, either the first or second lumbar puncture included in the study.
- Lidocaine Injection: Participants who received sham-EMLA cream (applied at least 60 minutes prior to procedure) and following conscious sedation, the patient received lidocaine 1% injection (~1-2ml) at the appropriate site 30-60 seconds prior to prior to procedure, either the first or second lumbar puncture included in the study.
Arm/Group | EMLA | Lidocaine Injection
Number analyzed (Participants) | 10 | 10
score on a scale
  Wong-Baker Faces Pain Rating Scale Score 30 - 60 minutes after waking up after lumbar puncture | 0 [0 to 0] | 0 [0 to 0]
  Wong-Baker Faces Pain Rating Scale Score 24 hours after lumbar puncture | 0 [0 to 8] | 0 [0 to 8]

2. Secondary Outcome: Post Lumbar Puncture PRN Pain Medication Usage
Description: Use of PRN or "as needed" pain medicine by the patient was determined. Patients with parent/guardian assistance were asked to record the "as needed" pain control medication, acetaminophen. the patient used within the 24 hours after lumber puncture. Counts of patients using acetaminophen in the 24 hours following lumber puncture are reported.
Time Frame: 24 hours following lumbar puncture
Measure: Count of Participants; unit: Participants
Groups:
- Lidocaine: Participants who received sham-EMLA cream (applied at least 60 minutes prior to procedure) and following conscious sedation, the patient received lidocaine 1% injection (~1-2ml) at the appropriate site 30-60 seconds prior to prior to procedure, either the first or second lumbar puncture included in the study.
Arm/Group | EMLA | Lidocaine
Number analyzed (Participants) | 10 | 10
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 7 days for each intervention
Arm/Group | EMLA | Lidocaine Injection
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT04003012/Prot_SAP_000.pdf